CLINICAL TRIAL: NCT01827397
Title: Phase 1 Randomised, Single-centre, Observer-blind, Placebo-controlled Trial of Safety and Immunogenicity of EN41-UGR7C HIV Vaccine Candidate Administered Intramuscularly in Healthy Female Volunteers
Brief Title: Safety & Immunogenicity of Immunisations With EN41-UGR7C HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PX'Therapeutics (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EN41CT1.1.2
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: - HIV
Keywords: Safety of this HIV vaccine
MeSH Terms: interventions — aluminum sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EN41-UGR7C HIV vaccine (Experimental): Group 1: IM injection of 210 µg UGR7-C in 560 µg of Alum at month 0, 1 and 4
  Interventions: Biological: EN41-UGR7C HIV vaccine
- NaCl (Placebo Comparator): Group 2: IM injection of 700 µL of 0.9% sodium chloride (NaCl) at month 0, 1 and 4
  Interventions: Biological: NaCl

INTERVENTIONS:
Biological: EN41-UGR7C HIV vaccine
  Other Names: EN41-UGR7C adjuvanted with Alum
  Arms: EN41-UGR7C HIV vaccine
Biological: NaCl
  Other Names: NaCl placebo vaccine
  Arms: NaCl

SUMMARY:
The purpose of the clinical trial is to evaluate the safety and immunogenicity in female volunteers of EN41-UGR7C vaccine candidate adjuvanted with Alum using IM administration. The objective of the immunisation is to induce mucosal and systemic binding and neutralizing antibodies against HIV in order to block the virus on the mucosal surface and neutralise the viral particles that may eventually succeed in crossing the mucosal barrier.

This is a Phase 1 exploratory study. EN41-UGR7C will be administered for the first time in humans.

Volunteers who are vaccinated with EN41-UGR7C may develop an immune response against HIV, but its ability to induce meaningful protection against HIV will not be known before Phase 3 efficacy trials are completed, as correlates of protection against HIV are not yet clearly defined.

Consequently, there is no direct benefit to volunteers. They will be reimbursed for their time and travel.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 18 and 55 years on the day of screening
2. Available for a maximal study duration of 8 months from screening
3. Willing and able to give written informed consent
4. At low risk of HIV infection and willing to remain so for the duration of the study defined as:

   * no history of injecting drug use in the previous ten years
   * no gonorrhoea or syphilis in the last six months
   * no high risk partner (e.g. injecting drug use, HIV infected sexual partner) either currently or within the past six months
   * no unprotected vaginal or anal intercourse in the last six months outside a relationship with a regular partner known to be HIV negative
   * no unprotected sex with someone from a high HIV prevalence region where HIV is more common than in the UK (e.g. Sub-Saharan Africa, Caribbean, South-East Asia)
5. Negative HIV1/2 antibody/antigen test result at screening
6. If heterosexually active female, using an effective method of contraception using a double barrier method of contraception (combined oral contraceptive pill, injectable or implanted contraceptive and use of condoms incorporating spermicide; physiological or anatomical sterility) from 14 days prior to the first vaccine administration until 3 months after the last administration, and willing to undergo urine pregnancy tests prior to each vaccine administration and blood pregnancy test at screening and final follow-up visits. Heterosexual females who become sexually active during the trial should also follow the same guidance
7. Agree to abstain from donating blood during their participation in the trial
8. Registered with a General Practitioner and medical history available for 12 months before dosing
9. Satisfactory response received from General Practitioner relating to medical history before randomization

Exclusion Criteria:

1. Pregnant or lactating or planning to get pregnant within the next year
2. Clinically relevant abnormality on history or examination:

   * central nervous system disorder or disease, including history of grand-mal epilepsy
   * severe eczema
   * clinically significant haematological, cardio-pulmonary, metabolic, gastrointestinal, renal, psychiatric or ophthalmological disorders
   * acute infection or illness
   * autoimmune disease, immunodeficiency or use of immunosuppressive agents in preceding 3 months prior to dosing
3. Known hypersensitivity to any component of the vaccine formulation used in this trial, or have severe or multiple allergies
4. History of severe local or general reaction to previous vaccination defined as:

   * local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
   * general: fever >39.5°C within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
5. Receipt of live attenuated vaccine within 60 days or other vaccine within 14 days of schedules study vaccine dosing
6. Receipt of an experimental vaccine containing HIV envelope proteins at any time in the past
7. Receipt of blood products or immunoglobulin within 4 months of screening
8. Participation in another trial of a medicinal product, completed less than 90 days prior to Visit 2 and planned participation in another clinical trial during the present trial
9. HIV 1/2 antibody/antigen positive or indeterminate on screening
10. Positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
11. Clinically significant abnormal result in routine laboratory parameters.
12. Unable to read and speak English to a fluency level adequate for the full comprehension of study and procedures required in participation and consent
13. Unlikely to comply with protocol
14. History of drug or alcohol abuse or regular use of drugs, or who test positive for alcohol test at screening
15. On regular medication which in the opinion of the investigator makes volunteer unsuitable for participation in the study
16. Any local vaginal, cervical or gynaecological condition which may interfere with collection or interpretation of data collected through vaginal samples
17. Using any Intra Uterine Contraceptive Device as there is a risk of dislodging, displacing or removing the device when pulling or removing Softcup used for vaginal sampling
18. Clinically significant abnormality on ECG performed at the screening visit
19. Any condition that, in the investigator's opinion, compromises the volunteer's ability to meet protocol requirements or to complete the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety of 3 EN41-UGR7C administrations | Up to 3 months after the last administration
  1. Safety assessed at any time from the first dose until 3 months after last administration by:Proportion of subjects developing Grade 3 or 4 adverse event
Assessment of EN41-UGR7C immunogenicity | Up to 3 months after the final administration
  Immunogenicity: to assess the EN41-UGR7C specific serum IgG responses measured by ELISA induced by the vaccine candidate up to 3 months after the final administration with a 3-fold increase from pre-administration baseline sample taken at visit 2, week 0.
  If no serum sample is available from this time point, serum taken at visit 1, screening, may be substituted.

SECONDARY OUTCOMES:
EN41-UGR7C specific ELISA IgA responses | Up to 3 months after the final administration
  -To measure the EN41-UGR7C specific ELISA IgA responses in serum and EN41-UGR7C IgA and IgG responses in vaginal samples up to 3 months after the final administration

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Johnson, Pr, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital; Royal Free London NHS Foundation Trust Pond Street, London, United Kingdom